CLINICAL TRIAL: NCT06213233
Title: Pragmatic Trial of Cannabidiol to Improve Chronic Pain Symptoms Among Veterans
Brief Title: MIVetsCan: Cannabidiol (CBD)-Care Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kevin Boehnke (Other)
Collaborators: Michigan, State of, Licensing and Regulatory Affairs (Unknown)
Responsible Party: Sponsor-Investigator, Kevin Boehnke, Research Assistant Professor, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM00231202; VMR2022-03 (Other: Michigan, State of, Licensing and Regulatory Affairs)
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Pain, Chronic
Keywords: Cannabidiol (CBD); Veterans; Surveys; Fitbit wearable
MeSH Terms: conditions — Chronic Pain | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cannabidiol (Experimental)
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Placebo — Participant will take placebo days 1-28 during study treatment. Given the pragmatic design, participants will be instructed to take the study drug whenever participants wish, with suggested starting dosing of 0.2 milliliter (mL) in the morning and 0.2mL in the evening (up to 1.2mL per day).
  Arms: Placebo
Drug: Cannabidiol — Participant will take Epidiolex days 1-28 during study treatment. Given the pragmatic design, participants will be instructed to take the study drug whenever participants wish, with suggested starting dosing of 0.2 milliliter (mL) in the morning and 0.2mL in the evening (up to 1.2mL per day).
  Other Names: Epidiolex
  Arms: Cannabidiol

SUMMARY:
This research is studying the effects of cannabidiol (CBD), an active component from cannabis (a.k.a. marijuana), on Veterans' chronic pain. The purpose of this study is to better understand if CBD can improve pain symptoms in Veterans with chronic pain.

Eligible participants will be randomly assigned to receive either placebo medication (not active) or CBD during the study period.

The study hypotheses:

- CBD would improve overall pain symptoms compared to placebo

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and speak English sufficiently to allow for written informed consent and patient-reported outcomes measures
* Armed Services Veteran
* All participants must have been enrolled in the MIVetsCan Pain Registry (HUM00223894) for at least 4 weeks and agree to continue participation in that study.
* Reports moderate to severe chronic pain defined by protocol
* Currently using or interested in using cannabis for pain management
* Self-reported willingness to refrain from or not increase current Tetrahydrocannabinol (THC) or other cannabis product use (including CBD) during the study intervention or other cannabinoid use during the study intervention
* Individuals of reproductive potential must agree to use acceptable birth control per protocol
* Participants must also agree not to donate sperm or eggs during study drug administration
* Willingness to attend all study visits (may be done virtually)
* Ability to take and to swallow the study medication and be willing to adhere to the treatment regimen
* Willingness to wear Fitbit or other similar sensor for passive-data collection
* Willingness to fill out daily diary via smartphone to assess symptom status, study drug use, and other cannabis use

Exclusion Criteria:

* Not an Armed Services Veteran
* Inability to provide informed consent (e.g., cognitive impairment, unable to sufficiently communicate in English)
* Participant reports pregnancy or are nursing
* Planning to move out of a state with legal recreational marijuana use during course of study
* Risk for imminent harm - Suicidal ideation or wish to die as assessed per protocol
* Any impairment, activity, behavior, or situation that in the judgment of the study team would prevent satisfactory completion of the study protocol
* Participation in any other clinical trials over the course of this study
* Medical or psychiatric conditions that in the judgment of study personnel would preclude participation in this study (e.g., psychosis, suicidal ideation; note that stable anxiety and depression are not exclusions)
* Having a serious or unstable hepatic disease (e.g., non-alcoholic fatty liver disease or liver cirrhosis)
* Individuals with major neurological disorders, such as dementia, Parkinson's disease, cognitive impairment, epilepsy, and seizures
* Recent/new diagnosis of cancer within the past 3 years (other than localized melanoma, localized basal cell carcinoma, localized squamous cell carcinoma treated or untreated)
* Current valproate and clobazam use per self-report or medical records
* Self-reported allergies to sesame oil or cannabis/cannabinoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Global impression of change (PGIC) between groups at end of treatment (Day 28) | Day 28
  This is a 1-item survey that measures patient perceptions of intervention success. This survey is scored from 1 to 7, where lower scores indicate a better outcome.

SECONDARY OUTCOMES:
Chronic pain severity between groups in the study period (Days 1 - 28) | Days 1-28
  Aggregated worst pain intensity (0-10 numerical rating scale) between groups during 7-day epochs from day 1 through day 28. Higher scores indicate worse pain.
Change in pain interference based on the pain interference 4a short form items from the Patient Reported Outcomes Measurement Information System (PROMIS)-29+2 Profile v2.1 | baseline (day 1), day 28
  There are 4-items on this survey that participants will complete regarding pain interference from not at all (1) - very much (5). Scores range from 4-20 with a higher score meaning more interference.
Anxiety based on the Patient Reported Outcomes Measurement Information System (PROMIS)-29+2 Profile v2.1 | Days 1-28
  There are 4-items on this survey that participants will complete regarding anxiety from never (1) - always (5). Scores range from 4-20 with a higher score meaning more anxiety.
Sleep disturbance based on the Patient Reported Outcomes Measurement Information System (PROMIS)-29+2 Profile v2.1 | Days 1-28
  This is a 4-item patient-reported scale indicating sleep quality. Scores range 4 to 20 with a higher score correspond to higher levels of sleep disturbance.
Change in suicidal ideation based on the Negative Suicide Ideation questionnaire (PANSI) | Baseline (day 1), 28
  The 8-items of vulnerability to suicidality participants will complete with answers from none of the time (1)-most of the time (5). Scores range from 8-40 with a lower score having fewer suicidal ideations.
Change in suicidal ideation based on Positive and Negative Suicide Ideation (PANSI) Inventory | Baseline (day 1), 28
  This is a 14-item subjectively completed inventory that consisted of 2 subscales: the PANSI-negative suicide ideation (NSI) subscale composed of 8 items and the positive ideation (PI) subscale consisting of 6 items. The possible total scores on the PANSI-NSI and PANSI-PI subscales range from 8 to 40 and 6 to 30, respectively. Higher scores on the PANSI-NSI and lower scores on the PANSI-PI reflect greater risk for suicidal behavior.
Safety assessed by the number of adverse events that are possibly, probably, or definitely related to the study drug between groups | Days 1-28
  Number of participants having the event, severity, expectedness, and relatedness to the study treatment. The study will utilize the Common Terminology Criteria for Adverse Events v.5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Boehnke, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bergmans RS, Wegryn-Jones R, Klida C, Kurtz V, Thomas L, Williams DA, Clauw DJ, Kidwell KM, Bohnert ASB, Boehnke KF. Protocol for a pragmatic trial of Cannabidiol (CBD) to improve chronic pain symptoms among United States Veterans. BMC Complement Med Ther. 2024 Jun 29;24(1):250. doi: 10.1186/s12906-024-04558-3. PMID 38951902